CLINICAL TRIAL: NCT04642274
Title: The Impact of ERAS Program in Cardiac Surgery on Patient Prognosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ERAS in CS
Record Dates: First submitted 2020-11-17; First posted 2020-11-24 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: ERAS
Keywords: ERAS; Cardiac surgery

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS (Experimental)
  Interventions: Other: Preoperative Strategies; Other: Intraoperative Strategies; Other: Postoperative Strategies
- Control (No Intervention)

INTERVENTIONS:
Other: Preoperative Strategies — Patient Education Preoperative Oral Carbohydrate Loading Nutritional Optimization Glycemic Control Anemia Correction Preoperative Hair Removal
  Arms: ERAS
Other: Intraoperative Strategies — Anesthetic Technique (Multimodal Analgesia) Antibiotics Glycemic Control Blood Transfusion Blood Conservation Optimization of Hemodynamics Protective Lung Ventilation Strategy Optimization of Anesthetic Depth Optimization of CPB Management
  Arms: ERAS
Other: Postoperative Strategies — Postoperative Analgesia Temperature Management Renal Protection Glycemic Control Early Extubation Early Oral Intake Maintain Drain Patency and Early Removal Early Ambulation Thromboprophylaxis
  Arms: ERAS

SUMMARY:
The aim of the study is to develop, verify and optimize the ERAS protocol for cardiac surgery.

DETAILED DESCRIPTION:
The aim of the study is to develop, verify and optimize the ERAS protocol for cardiac surgery, thereby improving the overall prognosis of cardiac surgery patients, reducing the incidence of complications, and shortening the length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years.
* Undergoing elective surgery.
* Scheduled for cardiac valve surgery with cardiopulmonary bypass.
* Body mass index (BMI) between 16.5 and 31 kg/m².
* American Society of Anesthesiologists (ASA) physical status classification of II or III.

Exclusion Criteria:

* Refusal to participate, refusal to sign the informed consent form, or inability to communicate.
* Participation in other clinical trials concurrently.
* Combined coronary artery bypass grafting or ascending aorta surgery.
* Emergency surgery.
* Active infective endocarditis.
* Previous history of cardiac surgery.
* Preoperative presence of neurocognitive disorders (NCD), depression, or other psychiatric conditions.
* Known abuse of alcohol, drugs, or anesthetics.
* Pregnant or breastfeeding women.
* Presence of other serious comorbidities that may impede enrollment or affect survival, such as malignancies or severe disabilities.

Termination of Intervention

Intervention will be terminated for the following reasons:

* Withdrawal of consent and request to exit the trial during the study period.
* Significant changes in surgical approach: including the addition of deep hypothermic circulatory arrest, intra-aortic balloon counterpulsation (IABP) support, extracorporeal membrane oxygenation (ECMO) support, etc.
* Medical necessity for termination of intervention, as determined by the investigator, for example: use of cardiopulmonary bypass more than twice during surgery; unexpected difficulties in weaning from cardiopulmonary bypass or extubation; continued treatment may pose a risk to the patient.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | Within 1 month after surgery

SECONDARY OUTCOMES:
Length of ICU stay | Within 1 month after surgery
Duration of mechanical ventilation after surgery | Within 1 week after surgery
Postoperative bowel motility | within 1 month after surgery
Overall hospitalization costs | Within 3 months after surgery
Transfusion requirements | within 1 month after surgery
Postoperative acute pain | within 1 month after surgery
  assessed using the Visual Analog Scale (VAS), ranging from 0 (no pain) to 10 (worst imaginable pain)
Quality of recovery | within 1 month after surgery
  assessed using the 15-item Quality of Recovery-15 (QoR-15) scale, with each item scored from 0 (very poor) to 10 (very good), for a total score of 150
Chronic pain | within 6 months after surgery
  Diagnostic Criteria of Chronic (postsurgical) Pain
  1. Chronic pain (persistent or recurrent for longer than 3 months) is present.
  2. The pain began or increased in intensity after surgery.
  3. The pain is in an area of preceding surgery.
  4. The pain persisted for at least 3 months after the initiating event.
  5. The pain is not better accounted for by an infection, a malignancy, a pre-existing pain condition or any other alternative
Patient's subjective comfort | within 6 months after surgery
  assessed using the Bruggrmann Comfort Scale (BCS)，it is a scoring tool for assessing patient comfort, ranging from 0 (persistent pain) to 4 (pain-free even when coughing)
Postoperative complications | within 6 months after surgery
  Including mortality and complications both in-hospital and post-discharge

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - The First Affiliated Hospital of AnHui Medical University, Hefei, Anhui
  - Ruijin Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Chest Hospital Affiliated to Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No